CLINICAL TRIAL: NCT05408286
Title: Impact of COVID-19 on Quality of Life After Hospital Discharge in Patients Treated With NIV/C-PAP: an Observational, Prospective Multicenter Study.
Brief Title: Post Covid-19 Quality of Life After Hospital Discharge in Patients Treated With NIV/C-PAP
Acronym: VIDI-CAP
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Principal Investigator, Bertolotti Marinella, biologa, Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria
Other Study IDs: VIDI
Record Dates: First submitted 2022-03-04; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- inclusion criteria: All patients aged ≥18 years admitted for COVID-19 pneumonia treated with NIV/CPAP, discharged to their home with a negative molecular swab and signed informed consent were included in the study.
  Interventions: Behavioral: administration of questionnaires

INTERVENTIONS:
Behavioral: administration of questionnaires — administration of questionnaires

SUMMARY:
A multicenter longitudinal study with data collection at 4 and 8 months after hospital discharge.

DETAILED DESCRIPTION:
The study population consisted of patients treated with NIV/CPAP, admitted to the COVID-19 wards of the AO SS Antonio e Biagio and Cesare Arrigo in Alessandria (the promoting center), the Azienda Sanitaria Locale Bt (Barletta, Andria, Trani) and the Azienda Socio Sanitaria Territoriale in Lecco, from November 2020 to June 2021. The study assessed at 4 and 8 months after hospital discharge in the patient's home environment, quality of life, residual disability, anxiety and insomnia.

Enrollment took place only after the approval of the Ethics Committee of each participating center.

ELIGIBILITY:
Inclusion Criteria:

All patients aged ≥18 years admitted for COVID-19 pneumonia treated with NIV/CPAP, discharged to their home with a negative molecular swab and signed informed consent were included in the study

Exclusion Criteria:

Exclusion criteria were set in; patients admitted for COVID-19 pneumonia treated with NIV/CPAP and invasive ventilation and patients with pre-existing cognitive disorders at the hospital admission date.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients treated with NIV/CPAP, admitted to the COVID-19 wards of the AO SS Antonio e Biagio and Cesare Arrigo in Alessandria (the promoting center), the Azienda Sanitaria Locale Bt (Barletta, Andria, Trani) and the Azienda Socio Sanitaria Territoriale in Lecco, from November 2020 to June 2021
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
COVID-19 qualità di vita | 8 mesi
  polmonite COVID-19 qualità di vita

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Bolgeo, PhD, Principal Investigator — Azienda Ospedaliera nazionale SS Antonio e Biagio e Cesare Arrigo, Alessandria, Italy, EU
Locations (1):
- Azienda ospedaliera nazionale SS Antonio e Biagio e Cesare Arrigo, Alessandria, Italy

IPD SHARING:
Plan to Share IPD: No